CLINICAL TRIAL: NCT00401869
Title: The Effect of PROCRIT on Hemoglobin and Hematocrit and the Relationship to Postoperative Function, Vigor and Strength in Patients Undergoing Primary Total Joint Arthroplasty: A Randomized, Parallel Group, Open-Label Trial
Brief Title: The Effect of PROCRIT (Epoetin Alfa) on Postoperative Vigor and Handgrip Strength (VIGOR Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho Biotech, Inc. (Industry)
Organization: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012205; NCT00526825 (obsolete NCT alias)
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Anemia
Keywords: vigor; function; well-being; hand-strength; surgery; anemia; transfusion; strength; quality-of-life
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study was to compare the effect of epoetin alfa to preoperative autologous blood donation (PAD) on postoperative vigor (a measure of functional ability and well-being) and handgrip strength in patients undergoing hip or knee surgery.

DETAILED DESCRIPTION:
Total joint arthroplasty (including hip and knee surgery) often leads to significant blood loss and may result in the need for blood transfusion. To prepare for this possibility, patients frequently donate their own blood in advance of their surgery so that it is available if transfusion is required during or after the procedure. This process of self-donation is known as preoperative autologous blood donation (PAD). PAD is associated with certain limitations including for example, worsening pre-operative anemia (potentially leading to the need for transfusion) and questionable cost-effectiveness. PROCRIT (Epoetin alfa) is a hormone that stimulates red blood cells production. Administration of PROCRIT (Epoetin alfa) is also used presurgically in anemic patients undergoing elective noncardiac, nonvascular surgery to increase hemoglobin levels (red blood cells) and reduce the need for transfusion during or after surgery. PROCRIT (Epoetin alfa) has been shown specifically to increase hemoglobin levels and reduce the need for blood transfusion in patients who undergo hip or knee surgery. However, no studies have been done to evaluate the ability of epoetin alfa to enhance energy and quality-of-life in patients having hip or knee surgery. This study was undertaken to compare two methods of blood management (Epoetin alfa treatment versus PAD) in terms of vigor score (functional activity and well-being). Other outcomes of study include handgrip strength, post-operative hemoglobin levels, and number of patients requiring transfusion. This was a randomized (patients were assigned to each treatment group by chance), open-label (both patient and physician know what treatment group the patient is assigned to) trial. Patients randomly assigned to treatment with PROCRIT (Epoetin alfa) received a subcutaneous injection of 600 IU/kg once weekly for 3 weeks preoperatively and then within 24 hours postoperatively. Patients in the PAD group were to donate 1 unit of blood before total knee arthroplasty, and 2 units of blood before total hip arthroplasty, as tolerated, beginning up to 28 days before surgery. Patients were not permitted to receive both study treatments. Daily oral iron supplementation was given in both treatment groups. It was recommended that blood transfusions should not be given if the patient had hemoglobin greater than or equal to 8 g/dL unless clinical symptoms or patient history warranted intervention. Investigators were instructed to use identical criteria for autologous and allogeneic blood transfusions. Baseline measurements including hemoglobin, hematocrit, red blood cell count, white blood cell count, reticulocytes, vigor, and handgrip strength were collected 28 to 21 days before surgery. Hemoglobin, vigor, and handgrip strength were repeated within 24 hours before surgery and again on Day 2, Day 4 or 5 (or discharge), and once between days 14 to 21 after surgery. Safety was assessed throughout the study by monitoring the occurrence and severity of adverse events including infection and thromboembolism. Patients assigned to the epoetin alfa group received 600 IU/kg PROCRIT (Epoetin alfa) administered subcutaneously (under the skin) once weekly for 3 weeks preoperatively and once 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective unilateral (one joint), primary total joint arthroplasty of hip or knee
* pretreatment hemoglobin level of 11 to 14 g/dL
* enrollment 21-60 days in advance of surgery

Exclusion Criteria:

* No uncontrolled hypertension
* No seizure disorder
* No history of deep vein thrombosis
* No significant gastrointestinal bleeding in previous 6 months
* No clinically significant hematologic, cardiovascular, neurological, pulmonary, endocrine, gastrointestinal, or genitourinary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 1999-02; Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
The change in VIGOR score (as assessed by questionnaire) from baseline to 1) within 24 hours of surgery; 2) post-op Day 2; 3) Day 4 or 5 or hospital discharge; and 4) between post-op days 14 and 21.

SECONDARY OUTCOMES:
Handgrip strength (JAMAR Hand Dynamometer using the stronger hand and in a standardized position and method repeated 3 times - the maximum force exerted was recorded), hemoglobin, and incidence of transfusion as described for primary outcome intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech, Inc. Clinical Trial, Study Director — Ortho Biotech, Inc.

REFERENCES:
- [Result] Keating EM, Callaghan JJ, Ranawat AS, Bhirangi K, Ranawat CS. A randomized, parallel-group, open-label trial of recombinant human erythropoietin vs preoperative autologous donation in primary total joint arthroplasty: effect on postoperative vigor and handgrip strength. J Arthroplasty. 2007 Apr;22(3):325-33. doi: 10.1016/j.arth.2006.11.002. PMID 17400086
- See also: Click here to view the journal abstract from the study manuscript. — http://download.veritasmedicine.com/PDF/CR005824_alimentarypharmacologyandtherapeutics.pdf